CLINICAL TRIAL: NCT02138331
Title: Phase 1 Study of The Effect of Cell-Free Cord Blood Derived Microvesicles On β-cell Mass in Type 1 Diabetes Mellitus (T1DM) Patients
Brief Title: Effect of Microvesicles and Exosomes Therapy on β-cell Mass in Type I Diabetes Mellitus (T1DM)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Wael Fouad Nassar, Senior Consultant of Nephrology., General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 666666; Cell Free MSC Exo
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Diabetes Mellitus Type 1; Microvesicles; Exosomes; Cord Blood; Mesenchymal Stem Cells
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exosomes (Experimental): The exosomes have exosome-associated proteins such as the tetraspanin proteins, CD9 and CD81, Alix, Tsg101, and RNA that consists primarily of short RNAs of less than 300 nm. Some of these RNAs are microRNAs that are predominantly pre-microRNAs..Additionally, CB-SC displayed very low immunogenicity as indicated by expression of a very low level of major histocompatibility complex (MHC) antigens and failure to stimulate the proliferation of allogeneic lymphocytes.
  Interventions: Biological: MSC exosomes.

INTERVENTIONS:
Biological: MSC exosomes. — Exosomes: (Size) 40-100 nm, (markers) CD63, CD9, Alix, TSG 101, HSP 70 Microvesicles: (Size) 100-1000 nm, (markers) Annexin V, Flotillin-2, selectin, integrin, CD40 metalloproteinase
  Other Names: Extacellular vesicles; Microvesicles

SUMMARY:
Type 1 diabetes mellitus is strictly autoimmune mediated disease destructing the islets β-cell of the pancreas. Mesenchymal stem cells and its microvesicles are reported as an anti-inflammatory agents. We hypothesis that intravenous infusion of cell free umbilical cord-blood derived MSC microvesicles may reduce the inflammatory state and hence improve the β-cell mass as well as the glycemic control of the patients of T1DM.

DETAILED DESCRIPTION:
* Twenty T1DM patients, age between 18-60 years with reduction of C-peptide chain more than 50%, C-peptide of more than 0.8 ng/mL at Screening and requiring insulin ≥0.4 IU per kg per day.
* Twenty T1DM patients of the same entry selection criteria will be subjected to all steps except the microvesicles administration as a control group.
* Study follow up period: Three months
* Gender: Both males and females are included
* Entry selection criteria include:

UACR less than 300, BUN between 10-20 mg/dl, serum creatinin between 0.6-1.4 mg/dl and normal liver enzymes, normal serum bilirubin, normal serum albumin and coagulation profile). C-peptide of more than 0.8 ng/mL at Screening. BMI 20-40 kgm/m2 - Exclusion criteria: Other autoimmune diseases. Pregnancy. Previous treatment with stem cells. All patients and controls will be investigated for HBV, HCV & HIV by PCR test before enrollment in the study and positivity for any of these parameters means exclusion of this patient from the study.

- The primary end point will be the end of three months follow up. At day (0):All patients and controls will be subjected to the following investigations: Liver functions tests, kidney functions tests, HbA1c, glucose tolerance test (GTT), fasting and 2 hrs.post prandial blood glucose levels, C-peptide chain level and calculated total daily insulin dose.

After three months (at the end of the study) the same investigations will be repeated.

Two intravenous infusions of cell free cord-blood derived mesenchymal stem cells [CB-MSC] microvesicles:

- The first dose will be purified exosomes, ranging between 40-180 nm, in a dose of the supernatant produced from (1.22-1.51) × 10 (6)/kg/IV.

(Characterization of exosomes:CD63, CD9, Alix, TSG 101, HSP 70).

- The second dose, after 7 days, will be the microvesicles, ranging between 180-1000 nm, in a dose of the supernatant produced from (1.22-1.51) × 10 (6)/kg/IV.

(Characterization of microvesicles: (Annexin V, Flotillin-2, selectin,integrin, CD40 metalloproteinase).

ELIGIBILITY:
Inclusion Criteria:

* UACR less than 300, BUN between 10-20 mg/dl, serum creatinin between 0.6-1.4 mg/dl and normal liver enzymes, normal serum bilirubin, normal serum albumin and coagulation profile). C-peptide more than 0.8 ng/mL at Screening. BMI 20-40 kgm/m2.

Exclusion Criteria:

* Other autoimmune diseases. Pregnancy. Previous treatment with stem cells. All patients and controls will be investigated for HBV, HCV & HIV by PCR test before enrollment in the study and positivity for any of these parameters means exclusion of this patient from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Total daily insulin dose | Three months
  All T1DM patients with identified pre-study insulin dose and exosomes and microvesicles will be given then weekly follow up of the total daily insulin dose will be measured. After 3 months We calculate the total daily dose of insulin that maintain the RBS levels between 120-160 mg/dl at any point of the evaluation period.

SECONDARY OUTCOMES:
Pancreatic β-cell Mass | 3 months
  Pancreatic β-cell Mass levels will be assessed before and after the 3 months study period of time.

OTHER OUTCOMES:
Hemoglobin A1c | Three months
  HbA1c levels before enrollment and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Nassar, MD, Study Chair — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Mervat El Ansary, MD, Study Director — Cairo University; Abdelnaser A Saad, MSc, Principal Investigator — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Mosaad A Hamid, MD, Principal Investigator — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Wael M Esa, MSc, Principal Investigator — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Sameh Shawki, MSc, Principal Investigator — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Marwa Mohammad, MSc, Principal Investigator — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Tamer Shehab, MRCP, Principal Investigator — Sahel Teaching Hospital, General Committee of teaching Hospitals and Institutes; Heba A Ghaffar, MSc, Principal Investigator — Cairo University
Locations (3):
- Egypt (3):
  - Sahel Teaching Hospital, Sahel, Cairo Governorate
  - Sahel Teaching Hospital - General Committee of Teaching Hospitals and Institutes, Shubrā, Cairo Governorate
  - Sahel Teaching Hospital, General Commettee of Teaching Hospitals and Institutes., Shubrā, Cairo Governorate

REFERENCES:
- [Result] Ezquer F, Ezquer M, Contador D, Ricca M, Simon V, Conget P. The antidiabetic effect of mesenchymal stem cells is unrelated to their transdifferentiation potential but to their capability to restore Th1/Th2 balance and to modify the pancreatic microenvironment. Stem Cells. 2012 Aug;30(8):1664-74. doi: 10.1002/stem.1132. PMID 22644660
- See also: doi:10.1186/1741-7015-10-3 Cite this article as: Zhao et al.: Reversal of type 1 diabetes via islet b cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Medicine 2012 10:3. — http://www.biomedcentral.com/1741-7015/10/3/prepub